CLINICAL TRIAL: NCT06203158
Title: Intestinal Epithelial Fucosylation Affects the Efficacy of Ustekinumab in Crohn's Disease
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2023-01-112
Record Dates: First submitted 2023-12-20; First posted 2024-01-12 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: IBD
Keywords: durg efficacy; Crohn's Disease; Ustekinumab; Intestinal Epithelial Fucosylation
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High fucosylation group: Immunohistochemistry was used to detect the fucosylation level in the intestinal tissue biopsy of patients with Crohn's disease at baseline. The fucosylation level in the baseline intestinal tissue was higher than 50% of the total.
- Low fucosylation group: Immunohistochemistry was used to detect the fucosylation level in the intestinal tissue biopsies of patients with Crohn's disease at baseline. The fucosylation level in the baseline intestinal tissue was less than 50% of the total.

SUMMARY:
The loss of response rate of ustekinumab(UST) is high, and the specific mechanism has not yet been elucidated. Molecular markers that can accurately predict the efficacy of UST are urgently needed to provide theoretical basis for guiding individualized treatment. Therefore, this study intends to explore the impact of intestinal epithelial fucosylation levels on the efficacy of UST in patients with Crohn's disease(CD), aiming to provide predictable molecular markers for UST to accurately treat CD.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with moderate to severe Crohn's disease
2. Receiving treatment with ustekinumab
3. Received colonoscopy and collected intestinal tissue samples before and after treatment

Exclusion Criteria:

1. Pregnancy
2. Hypersensitivity to any component of ustekinumab
3. Cognitive or developmental disabilities prevent you from completing this study
4. Combined with diseases such as RA, diabetes, systemic lupus erythematosus, intestinal tuberculosis, ischemic enteritis, radiation enteritis and tumors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inflammatory bowel disease (IBD) is a chronic inflammatory disease involving the digestive tract, including two clinical phenotypes: Crohn's disease (CD) and ulcerative colitis (UC).
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-12-26 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
clinical remission rate at 24 week | at 24 week
  A specialist will evaluate the HBI score at 24 week based on the patient's clinical symptoms and determine whether the patient is in clinical remission based on the score.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No